CLINICAL TRIAL: NCT02134522
Title: The Role of Obstructive Sleep Apnea in the Pathogenesis of Hepatic Steatosis in Obese Children and Adolescents
Brief Title: The Role of Obstructive Sleep Apnea in Children With Fatty Liver Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We were not able to recruit participants.
Sponsor: Yale University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1404013732
Record Dates: First submitted 2014-05-07; First posted 2014-05-09 (Estimated); Results first posted 2018-06-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Non Alcoholic Fatty Liver Disease
Keywords: non alcoholic fatty liver; childhood obesity; Sleep Apnea
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Pediatric Obesity; Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- C-PAP intervention (Experimental): Continuous positive airway pressure is a commonly prescribed therapy for obstructive sleep apnea which is recommended for the treatment of obstructive sleep apnea in children and adults.
  Interventions: Device: Continuous positive airway pressure (CPAP).

INTERVENTIONS:
Device: Continuous positive airway pressure (CPAP). — Continuous positive airway pressure is a commonly prescribed therapy for obstructive sleep apnea which is recommended for the treatment of obstructive sleep apnea in children and adults.
  Other Names: c-pap

SUMMARY:
The purpose of this study is to examine whether CPAP therapy can reduce or eliminate hepatic fat accumulation in obese children and adolescents.

DETAILED DESCRIPTION:
NAFLD is emerging as one of the most common complications of childhood obesity. It is associated with and predicts the metabolic syndrome, independent of overall obesity. Recently, studies in obese adolescents have demonstrated that increased ALT levels are associated with deterioration in insulin sensitivity and glucose tolerance, as well as with increasing FFA and triglyceride levels. Further studies showed that the prevalence of metabolic syndrome and prediabetes increases with the increases in hepatic fat content in a cohort of obese adolescents. Moreover, the investigators found that the fatty liver is associated with a pronounced dyslipidemic profile characterized by large VLDL, small dense LDL, and decreased large HDL concentrations. Fatty liver, independent of visceral and intramyocellular lipid content plays a central role in the impairment of liver, muscle and adipose insulin sensitivity in obese adolescents. Thus, fatty liver disease may be the hepatic component of the metabolic syndrome. The synthesis of triglycerides in the liver is nutritionally regulated, and its formation from simple carbohydrates requires multiple metabolic pathways, including glycolysis and pyruvate oxidation to generate acetyl-CoA for fatty acid synthesis, NADPH generation to supply the reductive power, packaging of fatty acids into a glycerophosphate backbone, and finally, lipoprotein packaging to export triglycerides. Recent studies have shown an association between fatty liver and obstructive sleep apnea (OSA), a condition that has been estimated to affect up to 27% of obese children. In particular, OSA has been associated with the ALT levels and with the degree of steatohepatitis. Despite those evidences and the importance of NAFLD in the development of metabolic diseases, the information concerning the association between fatty liver and OSA in obese children and adolescents is quite sparse and in particular is unclear whether OSA itself can cause NAFLD or the two conditions just coexist as obesity complications. In this study the investigators will test the hypothesis that OSA is one of the determinants of hepatic fat accumulation. To prove the investigators hypothesis the investigators will select a group of individuals with NAFLD and OSA, who will undergo a weight maintenance diet and Continuous Positive Airway Pressure (CPAP) for 12 weeks. CPAP is FDA approved and represents the leading therapy for obstructive sleep apnea in children over age 7 and 40 lbs. To evaluate the effect of the CPAP on the intra hepatic fat accumulation the investigators will evaluate hepatic fat content with MRI at baseline and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Sleep Apnea as diagnosed by clinical sleep study (Apnea Hypopnea index greater than 1)
* Evidence of NAFLD as diagnosed by screening MRI (hepatic fat fraction ≥5.5%) Obese child/adolescent between 9-21 years old
* Compliance with using C-pap as instructed

Exclusion Criteria:

* Medications or know disease known to alter glucose or insulin metabolism such as oral steroids, or certain psychiatric medications, such as Xeleca, Lithium and Paxil.
* Type 2 Diabetes Mellitus
* Medications for chronic anti-inflammatory effects
* Consumption of alcohol

Ages: 9 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Santoro, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- C-pap Intervention: Subjects who underwent measurement of the hepatic fat content before and after the C-pap
Period: Overall Study
Arm/Group | C-pap Intervention
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- C-pap Intervention: Subjects undergoing measurements of hepatic fat content before and after C-pap
Arm/Group | C-pap Intervention
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Gender: Female | 0
  Gender: Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Changes in Hepatic Fat Content
Description: Abdominal MRI to measure percent liver fat done at baseline and 12 weeks.
Time Frame: baseline and 12 weeks
Population: Presented is the change from baseline to 12 weeks in a single patient.
Measure: Number; unit: percentage of hepatic liver fat
Groups:
- C-pap Intervention: Subjects who underwent the measure of hepatic fat content before and after the C-pap
Arm/Group | C-pap Intervention
Number analyzed (Participants) | 1
percentage of hepatic liver fat | -4.8

2. Secondary Outcome: Changes in Two Hour Glucose
Description: 2 hour glucose measured by an oral glucose tolerance test done at baseline and 12 weeks. Data are presented as mg/dl.
Time Frame: baseline and 12 weeks
Measure: Number; unit: mg/dl
Arm/Group | C-pap Intervention
Number analyzed (Participants) | 1
mg/dl | 5

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | C-PAP Intervention
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-05-05): https://cdn.clinicaltrials.gov/large-docs/22/NCT02134522/Prot_SAP_000.pdf